CLINICAL TRIAL: NCT06318546
Title: Efficacy of Dexmedetomidine As Adjuvant to Intrathecal Bupivacaine in Decreasing Incidence of Post Spinal Shivering in Parturients Undergoing Caesarean Section
Brief Title: Dexmedetomidine in Spinal Anesthesia Decreasing Post Spinal Shivering in Caesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS59/2024
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-02

CONDITIONS: Post Spinal Shivering
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): This group will undergo spinal anesthesia using fentanyl (50 microgram) as adjuvant to intrathecal bupivacaine
  Interventions: Drug: Fentanyl
- Dexmedetomidine (Active Comparator): This group will undergo spinal anesthesia using dexmedetomidine (10mg) as adjuvant to intrathecal bupivacaine
  Interventions: Drug: Dexmedetomidine Injection [Precedex],,,

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex],,, — patients will receive 0.5ml (10 µg) Dexmedetomidine as an adjuvant to 2.2ml hyperbaric Bupivacaine hydrochloride 0.5%
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Fentanyl — will be given 0.5 ml of one ampoule (2ml) of 100µg fentanyl (Fentanyl Hameln® 0.1mg/2ml - Sunny pharm) equivalent to 25 µg fentanyl as an adjuvant to 2.2ml hyperbaric Bupivacaine hydrochloride 0.5%
  Arms: Control

SUMMARY:
The investigators will test the effects of intrathecal dexmedetomidine as adjuvant to intrathecal bupivacaine and it's direct effect in decreasing incidence of post spinal shivering in Parturients Undergoing Caesarean section

DETAILED DESCRIPTION:
A.Preoperative settings:

All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation. An informed written consent will be taken from every patient just before the surgery.

B.Intraoperative and postoperative settings:

On arrival to the operating room, baseline parameters such as ECG, mean arterial blood pressure, heart rate, and oxygen saturation will be recorded. Intravenous line will be inserted and IV Ringer's solution will be started, 500ml bolus will be given as a preload over 20 min before performing spinal anaesthesia and maintenance volume of 10ml\kg.

For each group, patients will be put in sitting position, the procedure will be performed under complete aseptic precautions, local anaesthesia will be administered by infiltration of the skin and subcutaneous tissues with 3-5 ml lidocaine 1% at L3-L4 and A 25-G needle will be used.

Both groups will be given 2.2ml {11-12 mg} hyperbaric Bupivacaine hydrochloride 0.5%

ELIGIBILITY:
Inclusion Criteria:

* • ASA I or ASA II patients Scheduled for CS under spinal anaesthesia.

  * Age 20-35 years.
  * Height ≤165 cm.
  * BMI ≤40.
  * Procedure duration ≤ 90 minutes.

Exclusion Criteria:

* • Patients with known neurologic and psychiatric illness.

  * Contraindications for spinal anaesthesia as patient refusal, bleeding or coagulation test abnormalities, local skin infection at spinal lumbar region, raised intracranial pressure and hypovolemia.
  * Spine abnormalities.
  * Systemic disorders like hematological, respiratory, cardiac, renal or hepatic insufficiency.
  * Allergy to any of the drugs used in the study.
  * Toxemia of pregnancy or hypertension with pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Post spinal shivering | From injection to 3 hours post operative
  will be observed following spinal anaesthesia and thereafter for 3 hours. It will be graded by a blinded observer during the intraoperative and postoperative period using the scale validated by Crossley and Mahajan [0 = no shivering, 1 = piloerection or peripheral vasoconstriction but no visible shivering, 2 = muscular activity in only one muscle group, 3 = muscular activity in more than one muscle group but not generalized shivering, 4 = shivering involving the whole body]. Grades 3, and 4 shivering for at least 3 min will be considered positive, and maximum shivering will be considered if generalized shivering interfering with ECG monitoring or ability of the mother to hold the baby. Positive shivering or lower grade shivering will be treated with an IV bolus of meperidine (0.5 mg/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Ragab, M.B.B.CH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All dana will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 1/2025
Access Criteria: Free